CLINICAL TRIAL: NCT06796517
Title: Risk Factor Analysis Study for the Efficacy Comparison Between Advanced Immunochemotherapy and Classical Immunochemotherapy: a Prospective Study for Relapsed/Refractory Lymphoma Patients
Brief Title: Immunotherapy in Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Sung-Soo Park (Other)
Collaborators: Yeouido St. Mary's Hospital (Other)
Responsible Party: Sponsor-Investigator, Sung-Soo Park, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: XC24OIDI0042; RS-2023-00216446 (Other Grant/Funding Number: Ministry of Food and Drug Safety)
Record Dates: First submitted 2025-01-19; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Relapsed/refractory High Grade B Cell Lymphoma; High Grade B-cell Lymphoma; Diffuse Large B Cell Lymphoma Relapsed; Primary Mediastinal Large B-Cell Lymphoma; Burkitt Lymphoma
Keywords: immunochemotherapy; B cell lymphoma; Relapsed; Refractory
MeSH Terms: conditions — Recurrence; Burkitt Lymphoma; Lymphoma, B-Cell | interventions — Immunotherapy, Adoptive; Antibodies, Bispecific; Immunoconjugates; Antibodies, Monoclonal; Proteasome Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum, Bone marrow
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Advanced immunochemotherapy: Relapsed/refractory high grade B cell lymphoma patients treated with either chimeric antigen receptor T cell therapy, bispecific antibody, or antibody-drug conjugate
  Interventions: Drug: CAR-T Therapy; Drug: Bispecific antibody; Drug: Antibody-Drug Conjugate
- Classical Immunochemotherapy: Relapsed/refractory high grade B cell lymphoma patients treated with either proteasome inhibitor, immune modulatory drug, or monoclonal antibody.
  Interventions: Drug: Monoclonal antibody; Drug: Proteasome Inhibitor; Drug: IMiD treatment

INTERVENTIONS:
Drug: CAR-T Therapy — It uses the patient's own T cells, and requires a manufacturing process to modify and expand T cells before infusion. It directly targets B cell specific antigens, such as CD19 or CD20.
  Groups: Advanced immunochemotherapy
Drug: Bispecific antibody — It uses a dual targeting mechanism to enhance specificity and immune activation. It is an off-the-shelf treatment, and doesn't require a manufacturing process of patient cells.
  Groups: Advanced immunochemotherapy
Drug: Antibody-Drug Conjugate — It is a targeted therapy consisting of a monoclonal antibody linked to a cytotoxic drug. The antibody binds to a specific antigen on cancer cells, delivering the cytotoxic agent directly to the tumor, minimizing systemic toxicity.
  Groups: Advanced immunochemotherapy
Drug: Monoclonal antibody — Monoclonal antibodies are lab-engineered antibodies that target specific antigens expressed on cancer cells. These commonly target CD20 (rituximab or obinutuzumab) to mediate immune destruction.
  Groups: Classical Immunochemotherapy
Drug: Proteasome Inhibitor — It blocks the activity of proteasomes, which role is degrading damaged proteins. This disruption induces apoptosis in cancer cells. Common agents include bortezomib and carfilzomib.
  Groups: Classical Immunochemotherapy
Drug: IMiD treatment — Immune modulatory drugs modulate the immune response by enhancing T-cell and NK cell activty to disrupt tumor progression. Common drugs include lenalidomide and thalidomide.
  Groups: Classical Immunochemotherapy

SUMMARY:
The goal of this observational study is to compare the efficacy of advanced immunochemotherapy and classical immunochemotherapy in relapsed/refractory high grade B cell lymophoma patients. The main question it aims to answer is:

Does advanced immunochemotherapy, including CAR-T therapy, bispecific antibody, and antibody-drug conjugate offer superior survival outcomes than when treated with classical immunochemotherapy, such as proteasome inhibitors, immune modulatory drugs, and monoclonal antibodies?

Researchers will compare patients receiving advanced immunochemotherapy with those receiving classical immunochemotherapy to determine if advanced therapies result in better survival outcomes.

Laboratory findings and electronic medical records (EMR) from participants will be used to assess survival outcomes and treatment-related safety profiles.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 to 74 years.
* Diagnosed with any of the following after January 2015: diffuse large B cell lymphoma, primary mediastinal large B cell lymphoma, high grade B cell lymphoma, or Burkitt lymphoma
* Patients who have received immunochemotherapy as treatment for relapsed/refractory lymphoma

Exclusion Criteria:

* Patients who have progressed to acute leukemia
* Patients who developed solid tumor during treatment
* Patients with active infectious status (acute pneumonia, viral infection, active hepatitis B state, or active pulmonary tuberculosis etc.)

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from Seoul St. Mary hospital and Yeoido St. Mary hospital
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the start of treatment or the date of study enrollment until death from any cause, assessed up to 100 months.
  Survival status is assessed through periodic follow-ups and medical records. Patients lost of follow-up are censored at their last known date of contact. The endpoint is either the date of death documented in medical records or the date of the last known follow-up for patients still alive.

SECONDARY OUTCOMES:
Progression-free survival | From the start of treatment or the date of study enrollment until disease progression or death from any cause, whichever comes first, assessed up to 100 months.
  Disease progression is determined based on clinical, radiographic, or laboratory data, using the Lugano criteria. Patients without documented progression at the time of analysis are censored at their last assessment date.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul St. Mary Hospital, Seoul
  - Yeoido St. Mary Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No